CLINICAL TRIAL: NCT01820988
Title: Cross-sectional Study on the Identification and Characterization of Community-dwelling Older People With Sarcopenia
Brief Title: MaSS - Maastricht Sarcopenia Study
Acronym: MaSS
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nutricia Research Fundation (Other)
Responsible Party: Sponsor
Other Study IDs: METC 13-3-006
Record Dates: First submitted 2013-03-12; First posted 2013-03-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sarcopenic vs. non-sarcopenic: Participants are classified as sarcopenic/non-sarcopenic according to the criteria of the European Working Group of Sarcopenia in Older People (EWGSOP).

SUMMARY:
The objective of this cross-sectional study is to obtain insight in the characteristics (nutritional status and level of physical activity) of sarcopenic compared to non-sarcopenic community-dwelling older people. There is one measurement moment and measurements will take place at the participant's home.

DETAILED DESCRIPTION:
* Characterization of sarcopenic older people (demographics, nutritional status, level of physical activity)
* Prevalence rates of sarcopenia in community-dwelling older people in the Netherlands
* Insight in differences and/or overlap between sarcopenia versus frailty
* Insight in the impact of sarcopenia on economic outcomes

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Have given informed consent
* Understand Dutch language
* Able to perform a walk test

Exclusion Criteria:

* Older people living in a nursing home
* Older people with active rheumatoid arthritis, post stroke status with evident lingering symptoms (paralysis, loss of motor functions), diseases of the nervous system like Parkinson and MS, active angina pectoris, dementia
* Older people in a wheelchair, with ICD or pacemaker

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older people
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean difference in nutritional status and level of physical activity of sarcopenic participants vs. non-sarcopenic participants, as a measure of a Food Frequency Questionnaire and Mini-Nutritional Assessment Tool and Minnesota questionnaire | 1 home visit

SECONDARY OUTCOMES:
Prevalence of sarcopenia in community-dwelling older people | 1 home visit
Number of sarcopenic participants with frailty as a measure of the FRAIL scale and Fried criteria | 1 home visit
Health care costs by sarcopenic vs. non-sarcopenic participants, measured by health care use | 1 home visit

CONTACTS AND LOCATIONS:
Overall Officials: J.M.G.A. Schols, Prof. Dr., Study Director — Maastricht University; R.J.G. Halfens, PhD, Principal Investigator — Maastricht University; J.M.M. Meijers, PhD, Principal Investigator — Maastricht University; D.M. Mijnarends, MSc, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Result] Mijnarends DM, Meijers JM, Halfens RJ, ter Borg S, Luiking YC, Verlaan S, Schoberer D, Cruz Jentoft AJ, van Loon LJ, Schols JM. Validity and reliability of tools to measure muscle mass, strength, and physical performance in community-dwelling older people: a systematic review. J Am Med Dir Assoc. 2013 Mar;14(3):170-8. doi: 10.1016/j.jamda.2012.10.009. Epub 2012 Dec 29. PMID 23276432
- [Result] Mijnarends DM, Schols JM, Meijers JM, Tan FE, Verlaan S, Luiking YC, Morley JE, Halfens RJ. Instruments to assess sarcopenia and physical frailty in older people living in a community (care) setting: similarities and discrepancies. J Am Med Dir Assoc. 2015 Apr;16(4):301-8. doi: 10.1016/j.jamda.2014.11.011. Epub 2014 Dec 17. PMID 25530211